CLINICAL TRIAL: NCT02729480
Title: Multi-center, Prospective, Controlled, Clinical Trial of Wireless CranioFacial Nerve Stimulation (CFNS) for the Treatment of CranioFacial Neuropathic Pain
Brief Title: Clinical Trial of Wireless CranioFacial Nerve Stimulation (CFNS) for the Treatment of CranioFacial Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Curonix LLC (Industry)
Collaborators: Goodman Campbell Brain and Spine, Indiana University, Indianapolis, Indiana, USA (Unknown); International Spine, Pain and Performance Center, Washington DC, USA (Unknown); Minimally Invasive Pain Institute, Utica, New York, USA (Unknown); Case Western Reserve University, Cleveland, Ohio, USA (Unknown); Pennsylvania Hospital, Philadelphia, Pennsylvania, USA (Unknown); Baylor College of Medicine (Other); Prizm Pain Management, Canton, Michigan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30-00208
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Facial Pain
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Continued Stimulation Group (Experimental): Subjects randomized to this group will have the Halo Craniofacial Nerve Stimulator System activated immediately.
  Interventions: Device: Halo Craniofacial Nerve Stimulator System
- Delayed Continuation Group (Active Comparator): Subjects randomized to this group with have the Halo Craniofacial Nerve Stimulator System activated after 90 days.
  Interventions: Device: Halo Craniofacial Nerve Stimulator System

INTERVENTIONS:
Device: Halo Craniofacial Nerve Stimulator System — The Halo Craniofacial Nerve Stimulator System is a wirelessly powered neurostimulator for pain in the face or head (not for headaches or migraine). This technology includes an implanted stimulator with an embedded receiver. The energy source is a small, external, rechargeable transmitter, which is worn by the patient. The transmitter sends the therapy program and power through the skin to the receiver.

SUMMARY:
The purpose of this study is to assess the effectiveness of craniofacial nerve stimulation for the treatment of neuropathic pain.

DETAILED DESCRIPTION:
Subjects will be randomized at enrollment into either a delayed or immediate continuation group. The immediate continuation group will immediately continue with the stimulation after a 30-day trial period and will be monitored for a total of 12 months. The delayed activation group will have their device turned off after the 30-day trial period for the next 3-months. At the 3-month visit, both groups be evaluated and the delayed activation group will have their devices reactivated.

Subjects will have neuropathic pain of various etiologies, including trauma, surgery or post-herpetic infections. Stimulators will be placed at the site target of the painful area, including the epifascial plane under the skin but above the muscles in the vicinity of the targeted branches of; A. Branches of Trigeminal Nerves in the Ophthalmic, Maxillary, or Mandibular B. Sensory branches of Facial Nerves C. Branches of the Occipital Nerves (Greater and/or Lesser) D. Branches of the Cervical Plexus (Superficial and/or Deep)

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age at time of informed consent
* Subjects have been diagnosed with Cranial-facial pain with an average VAS > 5 (on a 0-10 scale) over the course of the last month based on baseline pain diary.
* Subject diagnosis with neuropathic cranial-facial pain refractory to conventional medical management for at least 12 months prior to enrollment;
* Based on the medical opinion of the Principal Investigator, subject has a stable pain medication regimen for 3 months prior to study entry.
* Based on the medical opinion of the Principal Investigator, subject has a stable Tricyclic regimen for 3 months prior to study entry
* No medication overuse and not attributed to another causative disorder
* Based on the medical opinion of the Principal Investigator, there is no evidence of anatomic abnormalities that could jeopardize the placement of the device or pose a hazard to the subject;
* Based on the opinion of the Principal Investigator, subject is willing and able to operate the patient programmer, recharging equipment, diary and has the ability to undergo study assessments and provide accurate responses;
* Based on the opinion of the implanter, subject is a good surgical subject for the implant procedure;
* Subject is willing to undergo surgical implant procedure, attend visits as scheduled, and comply with the study requirements;
* Subject is male or non-pregnant female as determined with a negative pregnancy test at baseline visit, and if sexually active, must be using a medically acceptable method of contraception for the duration of their study participation;
* Subject is deemed to be neuro-psycho-socially appropriate for implantation therapies based of the assessment of a Clinical Psychologist, using face-to-face encounters and the psychological testing described in the measures;
* Patient is capable of giving informed consent

Exclusion Criteria:

* A. Subject has undergone botulinum toxin (BOTOX) injections of the head and/or neck in the last 3 months.
* Unresolved Malignancies in last six months;
* Subject has a history of migraine, headaches of central origin or trigeminal autonomic cephalalgias;
* Subject has postherpetic neuralgia (shingles);
* Complete deafferentation of all branches of the trigeminal, facial, occipital nerves and cervical plexus;
* Subject has an active systemic infection or is immune-compromised;
* Based on the medical opinion of the Principal Investigator, Psychologist and/or Psychiatrist, the subject has other psychological conditions (e.g., psychosis, suicidal ideation, borderline personality disorder, somatization, narcissism), other health conditions (e.g., substance abuse, another chronic condition requiring the regular use of opioid medication), or other legal concerns that would preclude his/her enrollment in the study or potentially confound the results of the study;
* Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study while participating in this study;
* Insulin-dependent diabetic who is not controlled through diet and/or medication (determined by the physician) or non-insulin dependent diabetic who is not well controlled through diet and/or medication;
* Bleeding complications or coagulopathy issues;
* Pregnant/lactating or not using adequate birth control;
* A life expectancy of less than one year;
* Any active implanted device whether turned off or on;
* A previous peripheral nerve stimulator (PNS) experience for the treatment of facial pain including a failed trial or explanted device;
* Conditions requiring Magnetic Resonance Imaging (MRI) evaluation or diathermy procedures;
* Subject is currently involved in litigation regarding injury, or is receiving worker's compensation benefits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Pain Score | 3 months
  To achieve a sustained 50% reduction in pain measured by the Visual Analog Scale (VAS)
Incidence and severity of adverse events | 3 months

SECONDARY OUTCOMES:
Percentage change from baseline in VAS for facial pain | Baseline and 3 months
Percent change from baseline in the Brief Pain Inventory-facial (BPIF) Questionnaire | Baseline and 3 months
Subject satisfaction with the therapy as measured by the Patient Global Impression of Change (PGIC) | 3 months
Change from baseline in quality of life, Physical component score using Medical Outcomes Short Form SF-36 | Baseline and 3 months
Change from baseline in quality of life, Mental component score using Medical Outcomes Short Form SF-36 | Baseline and 3 months
Change from baseline in pain rating index from the Short Form McGill Pain Questionnaire (MPQ-SF-2) | Baseline and 3 months

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - International Spine, Pain & Performance Center, Washington D.C., District of Columbia
  - Goodman Campbell Brain and Spine, Indiana University, Indianapolis, Indiana
  - Prizm Pain Management, Canton, Michigan
  - Minimally Invasive Pain Institute, Utica, New York
  - University Hospitals Case Medical Center, Department of Anesthesiology, Division of Pain Medicine, Cleveland, Ohio
  - Pennsylvania Hospital, Dept. of Neurosurgery, Philadelphia, Pennsylvania
  - baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for all primary endpoints will be made available within 6 months of study completion.